CLINICAL TRIAL: NCT02924519
Title: Postoperative Pain After Ambulatory Arthroscopic Shoulder Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Horsens (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-103-14
Record Dates: First submitted 2016-08-09; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Shoulder disorders are frequent, often associated with pain and occur in 7-34% of the general population and in 21% of the elderly population.

Of particular interest is prediction of postoperative pain after outpatient arthroscopic shoulder surgery since the clinical experience is that surgery does not always provides pain relief and the interindividual variation in acute postoperative pain intensity is significant. In addition, a Swedish study has shown that shoulder operations are associated with longer convalescence than other orthopaedic outpatient surgeries.

DETAILED DESCRIPTION:
This study is a prospective cohort with 6 months follow-up. Patients receive 5 questionnaires (preoperatively, 24 hours, 1 week, 3 months, 6 months, 1 and 2 years after surgery). The questionnaires contain questions about:

* Preoperative shoulder pain (type, intensity and duration)
* Preoperative pain in other areas besides the shoulder
* Brief Pain Inventory (BPI)
* Western Ontario Rotator Cuff Index (WORC)
* Single Assessment Numeric Evaluation (SANE)
* 3 validated physiological questionnaires:

  * State Trait Anxiety (STAI)
  * Pain Catastrophizing Scale (PCS)
  * Hospital Anxiety and Depression Scale (HADS)

In addition a cold pressor test is performed on the day of surgery to test the patients' threshold and ability to repress pain.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic shoulder surgery (subacromial decompression and acromioclavicular joint resection).

Exclusion Criteria:

* • < 18 years

  * mental disorders
  * Unable to speak and/or read Danish
  * Shoulder surgery within the last year
  * Raynauds phenomenon
  * Cuff suture
  * Biceps tenodesis
  * Labrum suture

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for ambulatory (outpatient) arthroscopic shoulder surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Chronic postoperative pain | 6 months after surgery
  Measured on a numerical rating scale (NRS; 0=no pain and 10=worst possible pain. Chronic postoperative pain is defined as NRS>=3 with an impact on daily living
Acute postoperative pain | 24 hours after surgery
  Measured on a numerical rating scale (NRS; 0=no pain and 10=worst possible pain. NRS>3= acute postoperative pain

SECONDARY OUTCOMES:
Acute postoperative pain | 1 week after surgery
  Measured on a numerical rating scale (NRS; 0=no pain and 10=worst possible pain. NRS>3= acute postoperative pain
Acute postoperative pain | 3 month after surgery
  Measured on a numerical rating scale (NRS; 0=no pain and 10=worst possible pain. NRS>3= acute postoperative pain
Preoperative psychological predictors for chronic pain | 6 months after surgery
  Hospital Anxiety and Depression Scale (HADS)
Preoperative psychological predictors for chronic pain | 6 months after surgery
  State-Trait Anxiety
Preoperative psychological predictors for chronic pain | 6 months after surgery
  Pain Catastrophizing Scale (PCS)
Preoperative physical predictors for chronic pain | 6 months after surgery
  Cold pressure test
Preoperative comorbidity | 6 months after surgery
  Other places than the shoulder

IPD SHARING:
Plan to Share IPD: No